CLINICAL TRIAL: NCT04516187
Title: Recognition of Serious Infections in the Elderly: Developing a Diagnostic Prediction Rule Based on Clinical Features and Blood Tests to Help Physicians Safely Rule Out a Serious Infection in an Older Patient Presenting to Ambulatory Care
Brief Title: Recognition of Serious Infections in the Elderly
Acronym: ROSIE
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Ann Van den Bruel, Professor, KU Leuven
Other Study IDs: S63771
Record Dates: First submitted 2020-07-30; First posted 2020-08-18 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Infection
Keywords: geriatric; diagnosis; ambulatory care; general practice; emergency care
MeSH Terms: conditions — Infections; Disease | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergency care: Consecutive enrolment of acutely ill older adults in emergency care
  Interventions: Diagnostic Test: signs and symptoms, blood tests
- General practice: Consecutive enrolment of acutely ill older adults in general practice
  Interventions: Diagnostic Test: signs and symptoms, blood tests

INTERVENTIONS:
Diagnostic Test: signs and symptoms, blood tests — signs and symptoms as observed by the treating physician + blood tests (CRP, Procalcitonin, White blood cell count)

SUMMARY:
The aim of this diagnostic accuracy study is to develop a clinical prediction rule based on signs, symptoms, patient characteristics and blood tests, to be used in ambulatory care to help physicians safely rule out a serious infection in an older patient.

It will be performed in general practices and emergency care departments across Flanders (Belgium).

DETAILED DESCRIPTION:
This is a cross-sectional diagnostic cohort study in older adults presenting to ambulatory care, including a follow-up period of 30 days. This study will be used to construct an algorithm consisting of clinical features and blood test results to identify serious infections.

The study will run in ambulatory care in Flanders. Recruitment is expected to last 2.5 years, with each patient entering the study only once. Older adults will be approached for possible participation in the study by practice staff. There is only one study visit.

Those who agree to participate via written informed consent will have demographics and clinical features recorded. A blood sample will be taken in all participants on study entry. Follow-up information for all participants will be collected using electronic medical record notes (EMD) and patient diaries.

Treatment and other management decisions will be left to the treating physicians' discretion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Presenting to a general practice with an acute illness with a maximum duration of 10 days since onset
* Suspicion of infectious disease (this may include suspicion of an acute exacerbation of COPD)
* Patient or proxy of the patient is willing and able to give informed consent for participation.

Exclusion Criteria:

The participant may not enter the study if any of the following apply:

* Too clinically unstable to waste time on study procedures
* Indwelling catheter in situ
* Immunocompromised or currently receiving medication for systemic immune-suppression, including corticosteroids
* Being admitted to hospital for longer than 24 hours less than 7 days before study entry, or having undergone surgery in the previous 30 days
* Living in a nursing home (both short term and long term stay) (only in general practice cohort)
* Patient was already included in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All acutely ill adults aged 65 years or older presenting to ambulatory care in whom a physician suspects an infection will be eligible. Ambulatory care is defined as in-hours general practice and emergency care.
Sampling Method: Non-Probability Sample
Enrollment: 493 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy 1 | 30 days
  Sensitivity and specificity of clinical prediction rules that are based on signs, symptoms, patient characteristics with and without blood tests, to be used in ambulatory care to help physicians safely rule out a serious infection in an older patient

SECONDARY OUTCOMES:
Diagnostic accuracy 2 | 30 days
  Sensitivity, specificity, positive and negative predictive value and likelihood ratios of individual signs, symptoms, patient characteristics and blood tests for diagnosing a serious infection in persons aged ≥65 years

OTHER OUTCOMES:
Net benefit: number of patients correctly classified as having a serious infection | 30 days
  To assess the added value of prediction model based decisions over treat all and treat none at clinically relevant thresholds
Diagnostic accuracy 3 | 30 days
  Sensitivity, specificity, positive and negative predictive value and likelihood ratios of tests across the most often occurring infection types
Descriptive 1: Prevalence (%) of serious infections in the study population | 30 days
  To investigate the potential for incorporation bias (diagnostic review bias) when establishing the reference standard in an expert review panel, with and without information on biomarker results.
Descriptive 2: multivariate analysis (no outcome) | 30 days
  To describe features independently associated with a physicians' gut feeling of serious infection in an older patient
Diagnostic accuracy 4 | 30 days
  Sensitivity and specificity of the developed prediction rules compared to existing prediction rules
Diagnostic accuracy, sensitivity analysis | 30 days
  Sensitivity and specificity of the prediction rules taking all-cause mortality versus mortality due to infection as an outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ann Van den Bruel, MD, PhD, Principal Investigator — Department of Public Health and Primary Care, KU leuven
Locations (12):
- Belgium (12):
  - De Driehoek Paal, Paal, Limburg
  - De Wijkpraktijk, Antwerp
  - De Leeuwenkaart, Brasschaat
  - Huisartsenpraktijk Arcade, Gelrode
  - De Bilter 28, Heers
  - Emergency Department Heilig Hart hospital Leuven, Leuven
  - Emergency Department University Hospitals Leuven, Leuven
  - Emergency Department St.-Jozef Hospital Malle, Malle
  - DRLA, Mortsel
  - De Driehoek Paal, Paal
  - Huisartspraktijk Brustempoort, Sint-Truiden
  - Onspraktijk, Wilrijk

IPD SHARING:
Plan to Share IPD: No